CLINICAL TRIAL: NCT06915597
Title: Procedural Success and Short- and Long-Term Outcomes of Drug-Coated Coronary Balloons Used in Different Clinical Scenarios
Brief Title: Drug-Coated Coronary Balloons in Different Clinical Scenarios
Acronym: DCB-DCS
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Pamukkale University (Other); Memorial Bahçelievler Hospital (Other); Bezmialem Vakif University (Other); Dicle University (Other); Ordu University (Other); Adana City Training and Research Hospital (Other); Marmara University (Other); Trakya University (Other); Kafkas University Health Research and Application Hospital (Unknown); Selcuk University (Other); Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Fatih Kahraman, Associate Professor, Kutahya Health Sciences University
Other Study IDs: DCB-DCS
Record Dates: First submitted 2025-03-19; First posted 2025-04-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: drug coted balloons; coronary artery disease; chronic total occlusions; de novo lesions; small vessel disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary artery disease: Patients with coronary artery disease who were treated with drug coated balloons will be included in the study.

SUMMARY:
Coronary stents are the best treatment method ever accepted in the treatment of coronary artery stenoses. Due to some limitations and complications of stent use, the operators tried to find new solutions. Drug Coated Balloons (DCBs) have been accepted as a new method in the treatment of in-stent restenosis and small vessel disease. Furthermore, they have been used in the treatment of de novo coronary lesions, chronic total occlusions and bifucation lesions. But data is limited in the short and long term success of DCBs in all these clinical scenarios. In our study we aimed to investigate the procedural success and short and long term outcomes of DCB use in different clinical scenarios.

DETAILED DESCRIPTION:
The DCB-DCS (Drug-Coated Balloon in Different Clinical Scenarios) Registry is a multicenter, observational study designed to evaluate the safety, feasibility, and clinical outcomes of drug-coated balloon (DCB) angioplasty in a broad spectrum of coronary artery disease presentations and lesion subsets in real-world practice across Türkiye. The registry aims to provide comprehensive evidence on contemporary DCB use beyond conventional in-stent restenosis, including de novo small and large vessels, bifurcation lesions, chronic total occlusions, acute coronary syndromes, and complex lesion morphologies.

Consecutive patients undergoing percutaneous coronary intervention (PCI) with a DCB-based strategy, either as a stand-alone therapy or in combination with bailout stenting, will be prospectively and retrospectively enrolled from participating high-volume centers. Detailed demographic, clinical, laboratory, angiographic, procedural, and pharmacological data will be systematically collected. Lesion characteristics will be classified according to standard angiographic and anatomical criteria, and procedural techniques including lesion preparation strategy (plain balloon, cutting/scoring balloon, high-pressure non-compliant balloon, atherectomy), use of intravascular imaging (IVUS, OCT, OFDI), and DCB type, size, and inflation protocol will be recorded.

The registry will assess short-term procedural success and long-term clinical outcomes, including major adverse cardiovascular events (MACE), target lesion failure, target vessel revascularization, myocardial infarction, stent thrombosis (when applicable), and all-cause and cardiovascular mortality. Subgroup analyses will explore the impact of different clinical presentations, lesion subsets, and procedural strategies on outcomes, with particular emphasis on the role of optimal lesion preparation, intravascular imaging guidance, and the need for bailout stenting.

By reflecting routine clinical practice in a large, unselected population, the DCB-DCS Registry seeks to define optimal procedural standards, identify predictors of success and failure, and generate hypothesis-forming data to guide future randomized controlled trials comparing DCB-based strategies with new-generation drug-eluting stents across diverse coronary scenarios.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years. Patients with coronary artery disease undergoing percutaneous coronary intervention (PCI) in whom a drug-coated balloon (DCB) is used as the intended treatment strategy for at least one target lesion.

DCB use in any clinical presentation, including stable coronary artery disease and acute coronary syndromes.

DCB treatment for different lesion subsets, including de novo lesions, in-stent restenosis, bifurcation lesions, small and large vessels, and chronic total occlusions.

Successful lesion preparation allowing DCB angioplasty (residual stenosis ≤30% and absence of flow-limiting dissection before DCB inflation, according to operator judgment).

Availability of baseline clinical, angiographic, and procedural data. Ability to provide informed consent for prospective enrollment or availability of data according to local regulations for retrospective inclusion.

Planned clinical follow-up.

Exclusion Criteria:

Primary treatment strategy without the use of a drug-coated balloon (e.g., exclusive drug-eluting stent implantation without DCB).

Cardiogenic shock at the time of index procedure. Life expectancy less than 1 year due to non-cardiac comorbidities. Contraindication to antiplatelet therapy. Known severe allergy to contrast media not amenable to premedication. Pregnancy. Inability to comply with clinical follow-up. Participation in another interventional clinical trial that could confound outcome assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (≥18 years) with coronary artery disease who undergo percutaneous coronary intervention (PCI) in routine clinical practice in participating centers and are treated with a drug-coated balloon (DCB) for at least one target coronary lesion. The registry will include patients across a broad spectrum of clinical presentations, including stable coronary artery disease and acute coronary syndromes, and will encompass a wide range of lesion subsets such as de novo lesions, in-stent restenosis, bifurcation lesions, small and large vessels, and chronic total occlusions. Both prospectively and retrospectively enrolled patients will be included, reflecting real-world practice without additional diagnostic or therapeutic interventions beyond standard of care. The population will therefore represent an unselected, all-comer cohort treated with contemporary DCB-based strategies, allowing comprehensive evaluation of clinical and procedural outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Death, target lesion revascularization, target vessel revascularization, myocardial infarction | 12 months
  Cardiac or noncardiac death events will be recorded during follow up. Forthermore, target vessel or lesion revascularization, myocardial infarction will be recorded according to the previously described criteria.

SECONDARY OUTCOMES:
Angina, target vessel revascularization, Procedural success and need for bailout stenting, Major bleeding (BARC ≥3) | 12 months
  Assessment of symptomatic angina status, need for repeat revascularization of the target vessel, procedural success including the requirement for bailout stent implantation, and the occurrence of major bleeding events defined as Bleeding Academic Research Consortium (BARC) type ≥3.

CONTACTS AND LOCATIONS:
Locations (5):
- Turkey (Türkiye) (5):
  - Pamukkale University, Denizli
  - Bahcelievler Memorial Hospital, Istanbul
  - Bezmialem Vakıf Universitesi, Istanbul
  - Goztepe Medicalpark Hastanesi, Istanbul
  - Kutahya City Hospital, Kütahya

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Aggregate data will be reported in publications and presentations. Access to patient-level data will be restricted to the study investigators in accordance with local regulations and data protection laws.